CLINICAL TRIAL: NCT02330575
Title: Alberta Cancer Exercise Community-based Program: A Pilot Randomized Controlled Trial
Brief Title: Alberta Cancer Exercise Pilot Randomized Trial
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); AHS Cancer Control Alberta (Other)
Responsible Party: Principal Investigator, Margie McNeely, Associate Professor, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA-CC-14-0153
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Participants in this group will receive standard education on the importance of physical activity in the recovery from cancer and how to become more active. Participants assigned to this group will have the option to participate in the exercise program after the 16-week follow-up assessment.
  Interventions: Behavioral: Education
- Supervised Community-based Exercise (Experimental): Participants in this group will take part in an 8-week supervised exercise program at the YMCA. Following the 8-week intervention, participants will have the option to continue for an additional 8-weeks at the YMCA (fee for service) or follow an 8-week self-directed program.
  Interventions: Behavioral: Exercise; Behavioral: Education

INTERVENTIONS:
Behavioral: Exercise — The participant exercise sessions will be conducted in small groups of 5 to 10 participants under the direct supervision of the community-based exercise specialist. Participants will have the choice between taking part in a bridging exercise class (e.g., Beauty program and Bridging to Fitness - Cancer) or group-based supervised fitness centre exercise training.
  Other Names: Physical Activity
  Arms: Supervised Community-based Exercise
Behavioral: Education — Participants allocated to the standard care group will receive standard advice and counseling on physical activity and will serve as the 'control group' for a 16-week period.

SUMMARY:
The purpose of the study is to examine the benefit and specific outcomes of a community-based exercise program that is designed to address the needs of individuals who are receiving or recovering from cancer treatment.

Eighty cancer survivors from Edmonton and Calgary will take part in the 24-week long study. Survivors will be randomly assigned to one of two groups. The first group will take part in an 8-week supervised exercise program followed by 8 weeks of self-directed or home-based exercise (early exercise group). The other 40 participants will continue with their normal activities for 16 weeks (delayed exercise group). After the 16 week period, participants in the delayed exercise group will take part in the 8-week supervised exercise program.

Exercise sessions will take place at selected YMCAs in Edmonton and Calgary. Exercise sessions will be supervised by specially trained exercise specialists who have received special training in exercise and cancer.

Outcomes of the study will include feasibility, physical fitness measures, cancer-related symptoms and quality of life.

DETAILED DESCRIPTION:
Purpose: The primary purpose of this proposed study is to pilot test the planned Alberta Cancer Exercise (ACE) program evaluation components at the level of the individual cancer survivor. These components include program reach as well as effectiveness as determined by outcomes of physical fitness, symptoms, and quality of life. This proposed study will enable us to formalize an evaluation strategy to inform effectiveness and implementation of the ACE program.

Methods: A randomized controlled trial (RCT) design will be utilized to examine the short-term effectiveness of the proposed community-based cancer exercise program designed for cancer survivors. The study will take place at the Cross Cancer Institute/University of Alberta and Tom Baker Cancer Centre/ University of Calgary as well as in selected YMCA community fitness centres in Edmonton and Calgary. The exercise intervention will be delivered by specially trained exercise professionals who have completed the formal cancer exercise education course. Eighty participants will be randomized to early (intervention group) or delayed community-based exercise programming (standard care group). Participants randomized to the intervention group will undertake the ACE Program at a selected Edmonton and Calgary YMCA for an 8-week period. Following the 8-week supervised intervention period, participants will have the option to continue on a 'fee for service' basis or to continue with self-directed exercise at home. Participants allocated to the standard care group will receive standard advice and counseling on physical activity and will serve as the 'control group' for a 16-week period. The standard care group will be offered participation in the 8-week ACE program at the completion of the 16-week follow-up period.

Outcomes: The primary outcome is program feasibility: recruitment, completion and adherence rates. For the purposes of the proposed study and the length of follow-up of 24 weeks, the RE-AIM components of Reach, Effectiveness and Implementation at the level of the individual will be evaluated as potential outcome indicators for the ACE program. Outcomes will include measures of health-related physical fitness, cancer-related symptoms and quality of life.

Summary: ACE is an active living initiative, encouraging cancer survivors in Alberta to take a role in their own wellbeing by supporting participation in cancer-specific community-based exercise programs.

ELIGIBILITY:
Inclusion Criteria:

1. Within 18 months of a diagnosis of any type of cancer
2. Receiving or have received curative cancer treatment (e.g., surgery, chemotherapy, radiation therapy)
3. Cleared for unrestricted physical activity by their treating oncologist

Exclusion Criteria:

1. Presence of metastatic disease
2. Any uncontrolled or serious comorbid conditions that would preclude participation in exercise testing and training
3. Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: number of participants completing the objective outcome measurements for the study | 24 weeks
  Proportion of subjects completing the physical fitness tests including aerobic capacity, musculoskeletal fitness and body composition measurements.

SECONDARY OUTCOMES:
Aerobic Capacity | 8 weeks
  Change in submaximal aerobic exercise capacity (treadmill, bike or 6 minute walk test)
Health-related Quality of Life | 8 weeks
  Change in quality of life: Functional Assessment of Cancer Therapy General Questionnaire
Symptom Assessment | 8 weeks
  Change in symptoms: Memorial Symptom Assessment Scale
Adherence to exercise | 24 weeks
  Attendance at supervised exercise sessions
Recruitment rate | 18 months
  Number of participants consenting to the study divided by the number of eligible participants
Upper Extremity Muscular Strength (optional) | 8 weeks
  Change in 8 repetition maximum strength of chest press
Upper Extremity Grip Strength (optional) | 8 weeks
  Hand Grip strength
Lower Extremity Muscular Strength (optional) | 8 weeks
  Change in 8 repetition maximum strength of leg press

OTHER OUTCOMES:
Adverse Events rate | 24 weeks
  Number of serious and minor adverse events
Program Costs | 24 months
  Costs related to study personnel, fitness centre costs and participant related costs
Body composition | 8 weeks
  Body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L McNeely, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary/ Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta/ Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
No plan in place